CLINICAL TRIAL: NCT07246694
Title: Combined Glossopharyngeal Nerve Block With Topical Anesthesia for Enhanced Recovery in Obstructive Sleep Apnea Patients Undergoing Uvulopalatoplasty
Brief Title: Enhanced Recovery After Uvulopalatoplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Uvulopalatoplasty Analgesia
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Analgesia; Recovery, Psychological
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): The patient will receive the ultrasound-guided glossopharyngeal nerve block combined with topical airway anesthesia.
  Interventions: Procedure: Glossopharyngeal nerve block
- Group c (Active Comparator): The patient will receive the standard multimodal analgesia.
  Interventions: Other: Standard multimodal analgesia

INTERVENTIONS:
Procedure: Glossopharyngeal nerve block — Glossopharyngeal nerve block using ultrasound guidance after induction of general anesthesia plus topical anesthesia before surgical incision.
  Arms: Group I
Other: Standard multimodal analgesia — The patient will receive intravenous fentanyl and non opioids analgesics (acetaminophen and non-steroidal anti-inflammatory drugs) with general anesthesia.
  Arms: Group c

SUMMARY:
Obstructive sleep apnea is a prevalent condition often treated surgically with palatoplasty, which improves airway patency and reduces apneic events. However, postoperative pain and airway discomfort following palatoplasty can be significant, leading to delayed oral intake, increased opioid consumption, and prolonged recovery. Combining an ultrasound-guided glossopharyngeal nerve block with topical airway anesthesia may provide synergistic analgesia and support a safer recovery profile.

DETAILED DESCRIPTION:
Obstructive sleep apnea is a prevalent condition often treated surgically with palatoplasty, which improves airway patency and reduces apneic events. However, postoperative pain and airway discomfort following palatoplasty can be significant, leading to delayed oral intake, increased opioid consumption, and prolonged recovery. Enhanced Recovery After Surgery protocols aim to accelerate functional recovery and reduce perioperative morbidity. Combining an ultrasound-guided glossopharyngeal nerve block with topical airway anesthesia may provide effective analgesia and support a smoother recovery profile.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of moderate to severe obstructive sleep apnea.
* Patients scheduled for elective palatoplasty under general anesthesia.
* American Society of Anesthesiologists Physical Status class I and II.

Exclusion Criteria:

* Patients with chronic opioid use.
* Advanced hepatic, renal, cardiovascular, and neurologic diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The recovery time | 1 hour
  The time from from inhalational anesthetic discontinuation to the first response to verbal command.

SECONDARY OUTCOMES:
Additional intraoperative analgesia | 4 hours
  Additional doses of intraoperative fentanyl.
Postoperative pain assessment | The first 24 hours postoperative.
  Postoperative pain assessment by the 10 points Visual Analogue Scale at at rest and during swallowing with 0 indicates no pain and 10 indicates the worst pain.
Total rescue analgesia | The first 24 hours postoperative.
  Total rescue analgesic dose needed during the first postoperative 24 hours.
Incidence of complications | 4 hours
  Incidence of any complications related to nerve block or local anesthesia such as hematoma formation or local anesthetic systemic toxicity.
Quality of recovery | The first 24 hours postoperative.
  Quality of recovery assessed by the Quality of recovery score-15 at the end of the first 24 hours postoperative. The Quality of recovery score ranges from 0 to150, with higher scores indicate better recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Mahmoud Ahmed, MD, Principal Investigator — Department of Anesthesia, Intensive Care & Pain Management, Zagazig University; Alshaimaa Abdelfattah Kamel, MD, Study Director — Department of Anesthesia, Intensive Care & Pain Management, Zagazig University; Osama Yehia Khalifa, MD, Study Director — Department of Anesthesia, Intensive Care & Pain Management, Zagazig University
Locations (1):
- Zagazig university hospital, Zagazig, Al-Sharkia, Egypt